CLINICAL TRIAL: NCT01811147
Title: Differentiating Unipolar and Bipolar Depression in Young Adults Using fMRI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB 12-1279
Record Dates: First submitted 2011-12-12; First posted 2013-03-14 (Estimated); Results first posted 2019-12-02 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Bipolar Disorder; Major Depression
Keywords: Bipolar; Depression; Mania; Hypomania; fMRI; antidepressant
MeSH Terms: conditions — Bipolar Disorder; Depressive Disorder, Major; Depression; Mania | interventions — Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (4):
- High Risk Depression (Experimental): Interventions will include the prescribing of Selective serotonin reuptake inhibitor or Serotonin-norepinephrine reuptake inhibitor antidepressants, bupropion or other antidepressant.
  Interventions: Drug: Selective Serotonin Reuptake Inhibitor (SSRI)
- Low Risk Depression (Experimental): Interventions will include the prescribing of Selective serotonin reuptake inhibitor or Serotonin-norepinephrine reuptake inhibitor antidepressants, bupropion or other antidepressant..
  Interventions: Drug: Selective Serotonin Reuptake Inhibitor (SSRI)
- Healthy Control (No Intervention): There is no intervention, but rather phone follow ups conducted as check ins to determine the continued eligibility of the healthy control participant.
- Bipolar (No Intervention): Bipolar participants are checked in with via phone conversations every three months, and have the opportunity to be scheduled for non-study visits to manage their symptoms.

INTERVENTIONS:
Drug: Selective Serotonin Reuptake Inhibitor (SSRI) — Subjects with depression will be treated with a Selective Serotonin Reuptake Inhibitor (SSRI) or a Serotonin-norepinephrine reuptake inhibitor (SNRI) for 24 months.
  Other Names: Serotonin-norepinephrine reuptake inhibitor
  Arms: High Risk Depression; Low Risk Depression

SUMMARY:
The purpose of the study is to find out what parts of the brain have increased or decreased activity and connectivity in individuals who have bipolar disorder, major depression, or no history of mood disorder. Another purpose of this study is to use MRI images to determine which young adults with major depression may be at greater risk for developing mild or more severe symptoms of mania which suggests a diagnosis of bipolar disorder.

DETAILED DESCRIPTION:
The study involves two phases, phase one includes the screening visit and MRI. The second phase, for depression participants, involves in person follow ups for up to two years. The second phase, for healthy and bipolar participants, involves phone follow ups, every three months for up to two years. The purpose of this study is listed above. We plan to enroll 200 participants total.

ELIGIBILITY:
INCLUSION CRITERIA FOR BIPOLAR DEPRESSED PATIENTS:

1. Ages 15 - 30 years (inclusive) and able to give voluntary informed consent (parents must also sign consent for subjects under 18)
2. Satisfy criteria for Diagnostic and Statistical Manual 4th edition (DSM-IV-TR) for Bipolar I or II disorder
3. Satisfy criteria for DSM-IV depressive episode-current
4. 17-item Hamilton Depression Rating Scale > 15 but < 25;
5. Young Mania Rating Scale score < 10
6. Satisfy criteria to undergo an MRI scan based on MRI screening questionnaire.
7. Able to be managed as outpatients during the study as ascertained by the following - i. Clinical Global Severity Scale < 5 i.e. moderately ill; ii. No significant suicidal or homicidal ideation or grossly disabled.

INCLUSION CRITERIA FOR ALL UNIPOLAR DEPRESSED PATIENTS:

1. Ages 15 - 30 years and able to give voluntary informed consent (Parental consent must also be obtained for those under 18 years old).
2. Satisfy criteria for DSM-IV-TR Major Depressive Episode using a Structured Interview
3. Never met criteria for mania or hypomania
4. 17-item Hamilton Depression Rating Scale score (HDRS) > 15 and < 25.
5. Young Mania Rating Scale (YMRS) score < 10
6. Satisfy safety criteria to undergo an MRI scan
7. Able to be managed as outpatients during the study as ascertained by the following - i. Clinical Global Severity Scale < 5 i.e. moderately ill; ii. No significant suicidal or homicidal ideation or grossly disabled

ADDITIONAL INCLUSION CRITERIA FOR HIGH RISK UD (HRUD) PATIENTS BESIDE THE INCLUSION CRITERIA FOR UD:

At least one of the following:

1. Family history of bipolar disorder in at least one first degree relative
2. History of any sub-threshold hypomania symptoms
3. History of mood episode related psychotic symptoms

ADDITIONAL INCLUSION CRITERIA FOR LOW RISK UD (HRUD) PATIENTS BESIDE THE INCLUSION CRITERIA FOR UD:

1. No family history of BD in a first or a second degree relative
2. No past history of any sub-threshold hypomania symptoms
3. No history of psychotic symptoms

EXCLUSION CRITERIA FOR DEPRESSION AND BIPOLAR SUBJECTS:

1. Meeting DSM-IV criteria for schizophrenia, schizophreniform disorder, schizoaffective disorder, mental retardation, pervasive developmental disorder.
2. History of receiving electroconvulsive therapy in the past 1 year
3. Use of neuroleptics, mood stabilizers or benzodiazepines in the past 2 weeks.
4. Use of antidepressants in the past 2 weeks.
5. If on fluoxetine in the past, then should not have been on this medication for 5 weeks.
6. Acutely suicidal or homicidal or requiring inpatient treatment.
7. Meeting DSM-IV criteria for other substance/alcohol dependence within the past 6 months or abuse in the past 3 months, excluding caffeine or nicotine. The criteria will be evaluated by interview and urinary toxicology screening. The use of caffeine or nicotine will be recorded.
8. Use of alcohol in the past 1 week before the MRI scan.
9. No serious acute or chronic medical or neurological illness, including previously known HIV positive status (due to possible CNS involvement) as assessed by history, physical examination and laboratory examination including EKG, CBC and blood chemistry.
10. Current pregnancy or breast feeding.
11. Metallic implants or other contraindication to MRI.

INCLUSION CRITERIA FOR HEALTHY CONTROLS: Healthy subjects matched for age, gender and ethnicity will be included

1. Ages 15 - 30 years (inclusive) and able to give voluntary informed consent (Parental consent must also be obtained for those under 18 years old)
2. No current or past history of psychiatric illness or substance abuse or dependence.
3. No current or past history of psychiatric illness or substance abuse or dependence in a first degree relative.

EXCLUSION CRITERIA FOR HEALTHY CONTROLS:

1. Pregnant or breast feeding.
2. Metallic implants or other contraindication to MRI.
3. Significant family history of psychiatric or neurological illness.
4. Currently taking any prescription or centrally acting medications.
5. Serious acute or chronic medical or neurological illness as assessed by history, physical examination and laboratory examination including CBC and blood chemistry.
6. Use of alcohol in the past 1 week and not being able to avoid alcohol use during the course of the study.

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 192 (Actual)
Dates: Start 2011-11; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Anand, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation Center for Behavioral Health, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Koirala P, Hu B, Altinay M, Li M, DiVita AL, Bryant KA, Karne HS, Fiedorowicz JG, Anand A. Sub-threshold bipolar disorder in medication-free young subjects with major depression: Clinical characteristics and antidepressant treatment response. J Psychiatr Res. 2019 Mar;110:1-8. doi: 10.1016/j.jpsychires.2018.12.006. Epub 2018 Dec 8. PMID 30579045

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After enrollment 3 subject were excluded form the study since it was later discovered that they did not meet the criteria.
Period: Overall Study
Arm/Group | High Risk Depression | Low Risk Depression | Healthy Control | Bipolar
Started | 51 | 56 | 49 | 33
Completed | 15 | 11 | 6 | 4
Not Completed | 36 | 45 | 43 | 29

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Risk Depression | Low Risk Depression | Healthy Control | Bipolar | Total
Number analyzed (Participants) | 51 | 56 | 49 | 33 | 189
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.67 (3.433) | 25.27 (3.661) | 24.24 (3.339) | 23.52 (3.784) | 23.99 (3.655)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 38 | 28 | 22 | 128
  Male | 11 | 18 | 21 | 11 | 61
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 37 | 50 | 37 | 26 | 150
  African American | 13 | 6 | 4 | 7 | 30
  Asian | 1 | 0 | 8 | 0 | 9
Region of Enrollment [Number; unit: participants]
  United States | 51 | 56 | 49 | 33 | 189

OUTCOME MEASURES:

1. Primary Outcome: HAM-D 17 Item: Hamilton Depression Rating Scale
Description: Hamilton depression rating scale (17-item HAM-D):
  Scores can range from 0 to 52: No depression (0-7); Mild depression (8-16); Moderate depression (17-23); and Severe depression (≥24).
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Risk Depression | Low Risk Depression | Healthy Control | Bipolar
Number analyzed (Participants) | 15 | 11 | 6 | 4
score on a scale | 6.6 (6.62) | 4.91 (4.11) | 2.333 (2.732) | 3.75 (4.992)

2. Secondary Outcome: YMRS: Young Mania Rating Scale
Description: Young Mania Rating Scale: Scores can range from 0 to 60: In Remission/No Mania (0-8); Mild (9-12); Moderate (13-18); Severe (19-25); Very Severe (>25)
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Risk Depression | Low Risk Depression | Healthy Control | Bipolar
Number analyzed (Participants) | 15 | 11 | 6 | 4
score on a scale | 0.2 (0.561) | 0 (0) | 0 (0) | 1.75 (3.5)

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | High Risk Depression | Low Risk Depression | Healthy Control | Bipolar
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/56 | 0/49 | 0/33
Serious Adverse Events (participants affected / at risk) | 5/51 | 3/56 | 0/49 | 0/33
Other Adverse Events (participants affected / at risk) | 3/51 | 4/56 | 0/49 | 0/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High Risk Depression (N=51) | Low Risk Depression (N=56) | Healthy Control (N=49) | Bipolar (N=33)
Sucidial Ideation (Psychiatric disorders) | 3 | 2 | 0 | 0
Hospitalization (Psychiatric disorders) | 1 | 1 | 0 | 0
Suicide Attempt (Psychiatric disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | High Risk Depression (N=51) | Low Risk Depression (N=56) | Healthy Control (N=49) | Bipolar (N=33)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 | 1 | 0 | 0
Visit to Emergency Room (Social circumstances) | 1 | 1 | 0 | 0
Substance Abuse Treatment (Psychiatric disorders) | 0 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol: Image Acquisition - CCF (2014-07-28): https://cdn.clinicaltrials.gov/large-docs/47/NCT01811147/Prot_000.pdf
  • Study Protocol and Statistical Analysis Plan: Full Protocol (2014-07-28): https://cdn.clinicaltrials.gov/large-docs/47/NCT01811147/Prot_SAP_001.pdf